CLINICAL TRIAL: NCT01783405
Title: Cardiovascular Disease in FH Heterozygous
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sociedad Española de Arteriosclerosis (Other)
Collaborators: Hospital Miguel Servet (Other); Universidad de Zaragoza (Other)
Responsible Party: Sponsor
Other Study IDs: D3560L00137
Record Dates: First submitted 2013-01-29; First posted 2013-02-04 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Familial Hypercholesterolemia
Keywords: LDLR mutation; Statin; Cardiovascular disease
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cases: FH heterozygous
- Controls: Parents of FH heterozygotes with FH

SUMMARY:
The objective of this project is to establish the current prevalence of cardiovascular disease in adult subjects suffering from genetically diagnosed HF, and to know the impact that drug treatment has course in cardiovascular disease when compared with that of their affected parents with a much longer period of exposure to hypercholesterolemia

DETAILED DESCRIPTION:
Familial hypercholesterolemia (FH) is the most common autosomal dominant disease in most countries, including Spain. Its prevalence is estimated at one in every 350-500 people being higher in certain areas with certain genetic isolation as French Canadians, Christian Lebanese, or "Afrikaners" in South Africa. The HF is characterized by a very high concentration of LDL cholesterol, familial autosomal dominant pattern, tendon xanthomas and increased risk of premature coronary disease. Without drug treatment, approximately 50% of men before age 50 years and the same percentage in women before age 60 will suffer a serious manifestation of cardiovascular disease. It has been estimated that HF limits life expectancy about 20 years for males and about 12 years for women, so that effective treatment is a priority in cardiovascular prevention. Most cases of HF are caused by mutations in the gene encoding the receptor of LDL particles (LDLR). More than 1000 different mutations in the LDLR gene (LDLR) have been described as the cause of HF, many of them specific to a territory or population group. In Spain we have described 235 different mutations and is one of the best studied populations in the world from the genetic point of view. This is because in Spain we have an efficient tool for genetic diagnosis of HF, referred Lipochip ® (Progenika Biopharma, Derio, Vizcaya), and allows us to be pioneers in the world in the diagnosis and treatment of HF.

Most cases of HF in Spain, and especially the cases with a genetic diagnosis, which represents the true diagnosis, are controlled by the Lipid Unit network of the Spanish Atherosclerosis Society (SEA) distributed throughout the national territory, and in many cases using homogeneous clinical criteria for the clinical management of these patients. For the above reasons the SEA is the ideal setting for studies in a wide range of subjects with HF, especially those requiring an accurate diagnosis. The advent of statins has been a landmark for people suffering from HF. Since the late 80s of last century we have this class of drugs. They have reduced and almost normalized LDL concentrations in FH and have substantively altered the natural progression of the disease. However, the health impact brought about by the statins in HF is unknown. Indirect data from the UK Simon Broome Register suggest that subjects with HF now have a better prognosis than 20 years ago but that register has many limitations that make difficult to know the real impact of the treatment.

Retrospective, obervacional, multicenter, based on Lipid Units of the Sociedad Española de Arteriosclerosis.

Our hypothesis is that statins have improved cardiovascular prognosis in recent years in heterozygous FH subjects. The objective of this project is to establish the current prevalence of cardiovascular disease in adult subjects suffering from genetically diagnosed HF, and to know the impact that drug treatment has course in cardiovascular disease when compared with that of their affected parents with a much longer period of exposure to hypercholesterolemia.

To establish the current prevalence of cardiovascular disease in adult subjects suffering from genetically diagnosed HF

To know the impact that drug treatment has resulted in cardiovascular disease when compared with that of their affected parents with a longer period of exposure to hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 30 and ≤ 70
* cLDL ≥ 95th percentile
* Functional mutation in LDLR or APOB in the proband or first degreee relative
* At least 10 years on statin treatment
* Lipid values and cardiovascular status of both parents

Exclusion Criteria:

* Same gender afected brothers of probands
* Homozygous FH

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heterozygous FH from the Lipid Units of the Sociedad Española de Arteriosclerosis (Spanish Atherosclerosis Society)
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Age first cardiovascular event | Baseline
  Age of first cardiovascular event is considered at the time of the last visit at the lipid clinic. Inclusion in the study has to be done within 6 moths from the last visit

SECONDARY OUTCOMES:
Age first stroke | Baseline
Age first coronary event | Baseline
Age first peripheral vascular disease | Baseline
Age diagnosis aortic aneurysm | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Civeira, MD, PhD, Principal Investigator — Universidad de Zaragoza
Locations (3):
- Spain (3):
  - Hospital San Jorge, Huesca
  - Hospital Universitario Miguel Servet, Zaragoza
  - Hospital Royo Villanova, Zaragoza